CLINICAL TRIAL: NCT04784715
Title: Phase III Study of Trastuzumab Deruxtecan (T-DXd) With or Without Pertuzumab Versus Taxane, Trastuzumab and Pertuzumab in HER2-positive, First-line Metastatic Breast Cancer (DESTINY-Breast09)
Brief Title: Trastuzumab Deruxtecan (T-DXd) With or Without Pertuzumab Versus Taxane, Trastuzumab and Pertuzumab in HER2-positive Metastatic Breast Cancer (DESTINY-Breast09)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D967UC00001; 2023-507904-30-00 (Registry Identifier: CTIS (EU)); 2020-004074-21 (EudraCT Number)
Record Dates: First submitted 2021-02-19; First posted 2021-03-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; HER2-positive; Metastatic
Keywords: Breast Neoplasms; Breast Diseases; Trastuzumab; Antineoplastic Agents, Phytogenic; Anti-drug conjugate; Molecular Mechanisms of Pharmacological Action;
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Breast Diseases | interventions — trastuzumab deruxtecan; taxane; pertuzumab; Trastuzumab

STUDY DESIGN:
Intervention Model Description: Study will consist of three arms:
  Arm A - trastuzumab deruxtecan with pertuzumab-matching placebo Arm B - trastuzumab deruxtecan with pertuzumab Arm C - standard of care (taxane [docetaxel or paclitaxel], trastuzumab and pertuzumab)
Masking Description: This study is open-label with respect to the control arm. Pertuzumab/placebo in the experimental arms will be blinded to the investigator and patients.
  The study will be "Sponsor-blind". To maintain the integrity of the study, Sponsor personnel directly involved in study conduct will not undertake or have access to efficacy data aggregated by treatment group prior to final data readout for the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Trastuzumab deruxtecan (T-DXd) plus pertuzumab-matching placebo
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Placebo
- Arm B (Experimental): Trastuzumab deruxtecan (T-DXd) plus pertuzumab
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Pertuzumab
- Arm C (Active Comparator): Standard of care (Taxane (paclitaxel or docetaxel), trastuzumab, and pertuzumab)
  Interventions: Drug: Taxane; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Administered by intravenous infusion
  Other Names: DS-8201a; T-DXd
  Arms: Arm A; Arm B
Drug: Placebo — Administered by intravenous infusion
  Arms: Arm A
Drug: Taxane — Investigator's choice of docetaxel or paclitaxel administered by intravenous infusion
  Arms: Arm C
Drug: Pertuzumab — Administered by intravenous infusion
  Arms: Arm B; Arm C
Drug: Trastuzumab — Administered by intravenous infusion
  Arms: Arm C

SUMMARY:
The study will evaluate the efficacy and safety of trastuzumab deruxtecan (also known as T-DXd, DS-8201a), either alone or in combination with pertuzumab, in treating patients with Human epidermal growth factor receptor 2 (HER2)-positive breast cancer as a first line of treatment in the metastatic setting.

DETAILED DESCRIPTION:
Eligible participants will be those diagnosed with HER2-positive (IHC 3+ or ISH+), metastatic breast cancer, who have received no prior chemotherapy or HER2-targeted therapy for advanced or metastatic breast cancer.

The study aims to evaluate the efficacy, and safety of trastuzumab deruxtecan, alone or with pertuzumab, compared with the standard of care treatment (taxane [docetaxel or paclitaxel], trastuzumab and pertuzumab). This study aims to see if trastuzumab deruxtecan allows patients to live longer without the cancer getting worse, or simply to live longer, compared to patients receiving standard of care chemotherapy. This study is also looking to see how the treatment and the cancer affects patients' quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be ≥18 years of age
* Pathologically documented breast cancer that:

  1. is advanced or metastatic
  2. is locally assessed and prospectively centrally confirmed as HER2-positive (IHC3+ or ISH+)
  3. is documented by local testing as hormone receptor (HR)-positive or HR-negative disease in the metastatic setting
* No prior chemotherapy or HER2-targeted therapy for advanced or metastatic breast cancer or only 1 previous line of endocrine therapy in the metastatic setting. Participants who have received chemotherapy or HER2-targeted therapy in the neo-adjuvant or adjuvant setting are eligible if > 6 months from treatment to metastatic diagnosis.
* Has protocol-defined adequate organ and bone marrow function
* ECOG performance status 0 or 1

Key Exclusion Criteria:

* Ineligible for any of the agents on the study.
* Any substance abuse or other medical conditions that, in the investigator's opinion, may interfere with subject's participation or study results
* Patients with spinal cord compression or clinically active central nervous system metastases. Participants with clinically inactive brain metastases or treated brain metastases that are no longer symptomatic may be included in the study.
* Active or prior documented interstitial lung disease (ILD)/pneumonitis or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Prior randomization or treatment in a previous trastuzumab deruxtecan study regardless of treatment arm assignment

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1157 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) assessment | Until progression or death, assessed up to approximately 60 months
  Defined as time from date of randomisation until the date of objective radiological disease progression according to Blinded Independent Central Review (BICR) using RECIST 1.1 or death by any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by Investigator assessment | Until progression or death, assessed up to approximately 60 months
  Defined as time from date of randomisation until the date of objective radiological disease progression according to Investigator using RECIST 1.1 or death by any cause.
Overall Survival (OS) | Until death, assessed up to approximately 104 months
  OS is defined as the time from randomisation until the date of death due to any cause.
Objective Response Rate (ORR) by BICR and Investigator assessment | Until progression or death (in the absence of progression), assessed up to approximately 60 months
  ORR is defined as The proportion of participants who have a complete response (CR) or partial response (PR) based on BICR and investigator assessment using RECIST 1.1.
Duration of Response (DoR) by BICR and Investigator Assessment | Until progression or death (in the absence of progression), assessed up to approximately 60 months
  DoR is defined as the time from date of first detection of objective response until the date of objective radiological disease progression according to BICR and investigator assessment using RECIST 1.1 or death in the absence of progression.
Time to second progression or death (PFS2) by Investigator assessment | Assessed up to approximately 104 months
  PFS2 is defined as the time from randomisation until the date of tumor progression on next-line treatment (the earliest of the progression event subsequent to first subsequent anticancer therapy after the first progression) or death from any cause; second progression will be defined according to local standard clinical practice.
To assess the effect of T-DXd ± pertuzumab relative to THP in terms of patient-reported pain in participants with HER2 positive, first-line mBC'. | Assessed up to approximately 60 months
  Pain progression: Time to sustained deterioration of European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 Pain Scale. Scores range from 0-100 based on 2 items with responses ranging from 1-4. A lower score would mean better outcome.
To assess patient-reported treatment tolerability | Assessed up to approximately 60 months
  Proportion of participants experiencing treatment related symptoms as measured by selected items from the European Organisation for Research and Treatment of Cancer, general cancer module (EORTC QLQ-C30), score of 1-4. A lower score would mean better outcome.
To assess patient-reported treatment tolerability | Assessed up to approximately 60 months
  Proportion of patients reporting different levels of overall tolerability as measured by the Patient Global Impression of Treatment Tolerability (PGI-TT), score of 0-4. A lower score would mean a better outcome.
To assess patient-reported treatment tolerability | Assessed up to approximately 60 months
  Proportion of participants experiencing treatment related symptoms as measured by selected items from the European Organisation for Research and Treatment of Cancer, breast cancer module (EORTC QLQ-BR45), score of 1-4. A lower score would mean better outcome.
To assess patient-reported treatment tolerability | Assessed up to approximately 60 months
  Proportion of participants experiencing treatment related symptoms as measured by selected items from the Patient-Reported Outcomes- Common Terminology Criteria for Adverse Events (PRO-CTCAE). PRO-CTCAE responses are scored from 0 to 4 (or 0/1 for absent/present). A lower score would mean a better outcome.
To assess patient-reported treatment tolerability | Assessed up to approximately 60 months
  The proportion of participants with maintained or improved physical function while on treatment, based on the EORTC QLQ-C30 Physical Functioning scale. Scores range from 0-100, based on 5 items with responses ranging from 1-4. A higher score would mean a better outcome.
Serum concentration of trastuzumab deruxtecan and pertuzumab | Up to Cycle 6, approximately Week 18; each cycle is 21 days
  Determination of trastuzumab deruxtecan and pertuzumab concentrations in serum.
Immunogenicity of trastuzumab deruxtecan. | Up to follow-up period, approximately 60 months
  Number and percentage of participants who develop anti-drug antibody (ADA) for trastuzumab deruxtecan.
Safety and tolerability of trastuzumab deruxtecan, alone or with pertuzumab | Assessed up to approximately 60 months
  Number of AEs according to NCI-CTCAE Version 5.0 per each treatment arm

CONTACTS AND LOCATIONS:
Locations (230):
- United States (28):
  - Research Site, Tucson, Arizona
  - Research Site, Springdale, Arkansas
  - Research Site, Glendale, California
  - Research Site, Longmont, Colorado
  - Research Site, Miami, Florida
  - Research Site, Palm Bay, Florida
  - Research Site, Plantation, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Louisville, Kentucky
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Summit, New Jersey
  - Research Site, New York, New York
  - Research Site, Shirley, New York
  - Research Site, York, Pennsylvania
  - Research Site, Germantown, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Denton, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Shenandoah, Texas
  - Research Site, Tyler, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Tacoma, Washington
- Argentina (10):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Caba
  - Research Site, Capital Federal
  - Research Site, Cipolletti
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Salvador de Jujuy
- Belgium (7):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
- Brazil (9):
  - Research Site, Florianópolis
  - Research Site, Goiânia
  - Research Site, Londrina
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
  - Research Site, Sorocaba
  - Research Site, Vitória
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Ste-Foy, Quebec
  - Research Site, Saskatoon, Saskatchewan
- China (22):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
- Denmark (3):
  - Research Site, Copenhagen O
  - Research Site, Sønderborg
  - Research Site, Vejle
- France (14):
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Le Mans
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (11):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Münster
  - Research Site, Paderborn
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Szolnok
- India (8):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Calicut
  - Research Site, Gūrgaon
  - Research Site, Mysuru
  - Research Site, Nashik
  - Research Site, New Delhi
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (9):
  - Research Site, Bergamo
  - Research Site, Candiolo
  - Research Site, Genova
  - Research Site, Livorno
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Rozzano
  - Research Site, Udine
- Japan (29):
  - Research Site, Akashi-shi
  - Research Site, Aomori
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukushima
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kawasaki-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Tsu
  - Research Site, Yokohama
- Mexico (6):
  - Research Site, Alc. Cuauhtémoc
  - Research Site, Estado de México
  - Research Site, Guadalajara
  - Research Site, Metepec
  - Research Site, Nuevo León
  - Research Site, Veracruz
- Peru (2):
  - Research Site, Arequipa
  - Research Site, Lima
- Philippines (7):
  - Research Site, Baguio City
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Quezon City
  - Research Site, San Juan City
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Floreşti
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- South Africa (7):
  - Research Site, Cape Town
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
  - Research Site, Rondebosch
  - Research Site, Soweto
- South Korea (4):
  - Research Site, Cheonan-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (5):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Vaxjo
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Karşıyaka
  - Research Site, Malatya
  - Research Site, Samsun
- United Kingdom (7):
  - Research Site, Buckhurst Hill
  - Research Site, Edinburgh
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Swansea
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tolaney SM, Jiang Z, Zhang Q, Barroso-Sousa R, Park YH, Rimawi MF, Saura C, Schneeweiss A, Toi M, Chae YS, Kemal Y, Chaudhari M, Sendur MAN, Yamashita T, Casalnuovo M, Danso MA, Liu J, Shetty J, Herbolsheimer P, Loibl S; DESTINY-Breast09 Trial Investigators. Trastuzumab Deruxtecan plus Pertuzumab for HER2-Positive Metastatic Breast Cancer. N Engl J Med. 2025 Oct 29. doi: 10.1056/NEJMoa2508668. Online ahead of print. PMID 41160818
- See also: BreastCancerStudyLocator.com — https://breastcancerstudylocator.com/
- See also: Daiichi Sankyo Contact for Clinical Trial Information Phone: 908-992-6400 — http://CTRinfo@dsi.com